CLINICAL TRIAL: NCT06534008
Title: The Effect of Combined Aerobic and Muscle Strengthening Exercises on Structural and Functional Cardiovascular Adaptations in Endometrial Cancer Survivors
Brief Title: Strive Cardio for Endometrial Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jess S. Gorzelitz (Other)
Responsible Party: Sponsor-Investigator, Jess S. Gorzelitz, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202311588
Record Dates: First submitted 2024-07-12; First posted 2024-08-01 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-07

CONDITIONS: Endometrial Cancer; Cardiovascular Diseases
Keywords: Functional Fitness; Arterial stiffness; Health Behaviors; Home-based; Exercise; Muscle Strengthening; Aerobic Endurance; Flexibility; Agility; Telehealth; Strength
MeSH Terms: conditions — Endometrial Neoplasms; Cardiovascular Diseases; Health Behavior; Motor Activity

STUDY DESIGN:
Masking Description: Outcomes assessor will be blinded to exercise status of participant but all participants will receive treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 12-week Exercise Intervention (Experimental): In this single-arm study, every participant will be enrolled in the 12-week distance-based exercise intervention. All participants will receive an exercise regimen and the necessary materials to complete and measure their exercise. All participants will receive weekly online heath coaching.
  Interventions: Behavioral: 12-week home-based exercise intervention

INTERVENTIONS:
Behavioral: 12-week home-based exercise intervention — All participants will be given the same 12-week distance-based exercise intervention.

SUMMARY:
STRIVE Cardio is a 12-week exercise intervention study with the goal to improve functional fitness and cardiovascular health for women who have completed treatment for non-metastatic endometrial cancer within the last five years and are currently in remission. Measures will include a functional fitness test, carotid-femoral pulse wave velocity, brachial artery flow mediated dilation, and a blood draw. Participants will be provided resistance bands, a dumbbell, and a Fitbit to keep. Participants will be compensated $50 for each of their two in-person visits.

DETAILED DESCRIPTION:
STRIVE Cardio is a distance-based exercise study for women who have completed treatment for non-metastatic endometrial cancer within the last five years and are currently in remission.

The intervention itself is 12 weeks of exercise, with one week of accelerometer wear prior to exercise with an additional week to schedule post-study visit procedures, yielding a total intervention length of 14 weeks. The exercise intervention will consist of (a) in-person pre-intervention study measures; (b) instructional materials (e.g. detailed exercise manual) and exercise training equipment (e.g. resistance bands, adjustable dumbbell, Fitbit Charge 5); (c) a virtually delivered instructional session; (d) access to informational web materials; (e) Support and feedback provided via virtual health coaching sessions; and (f) in-person post-intervention study measures.

Health coaching sessions will be delivered virtually and consist of (a) an initial health coaching session during week one discussing the participant's visions for health and wellness and overall goals of completing the intervention exercises; (b) sessions delivered once per week through week four discussing progress, barriers, facilitators, self-efficacy, and motivations for exercise goals to facilitate exercise adoption; (c) a midpoint check-in including a non-bias report from their health coach describing their progress thus far in the intervention. Participants then have the personal option to continue meeting with their health coach on a weekly basis or taper their health coaching sessions to include only weeks eight and eleven; (d) a final in person health coaching session to conclude.

The investigator's primary objective is to measure changes biomarkers of vascular structure and function following combined aerobic and muscle strengthening exercise in endometrial cancer survivors. The investigators hypothesize that there will be clinically meaningful improvements in structural and functional vascular biomarkers, and improved composite risk scores.

The investigator's two aims are to (1) Quantify the changes in vascular structure (pulse wave velocity) and function (flow mediated dilation) following a distance-based exercise program; and (2) Determine the magnitude of changes in ASCVD risk profiles following a distance-based exercise program.

ELIGIBILITY:
Inclusion Criteria

* Willing and able to provide written informed consent
* Willing to comply with study procedures and available for the duration of the study
* Fluent in spoken and written English
* Women 18 years of age or older
* Documented diagnosis of Type I, stage I-IIIc endometrial cancer within the past 5 years
* Completion of current cytotoxic treatment for endometrial cancer
* Technology access (phone call access, broadband internet, Wi-Fi) for tele coaching
* Comfort and willingness to use technology (videoconferencing) throughout the study for coaching
* Pass the Physical Activity Readiness Questionnaire (PAR-Q)
* Medical clearances given by their primary provider / oncologist (if indicated by the PAR-Q)

Exclusion Criteria

* Absolute contraindications to exercise (i.e., acute myocardial infarction, severe orthopedic or musculoskeletal limitations)
* History of previous myocardial infarction, ischemia, or hemorrhagic stroke
* Medically documented history of heart disease including heart valve disease, coronary artery disease, heart failure, peripheral artery disease, aortic disease, pericardial disease, cerebrovascular disease, or deep vein thrombosis
* Medical documentation of treatment-resistant hypertension OR taking ≥2 medications to treat hypertension
* Medically documented history of cardiovascular disease including (but not limited to): bypass surgery, stent procedures, bypass grafts, or coronary angioplasty
* Medically documented or self-reported type 1 diabetes (insulin-dependents)
* Prescriptions for or use of semaglutide (GLP-1 agonists) including name brands: Ozempic, Wegovy or Mounjaro
* Current or recent (within last 3 months) use of hormone replacement therapy (HRT)
* Evidence of recurrent or metastatic disease
* Currently performing resistance training ≥2 days per week
* Currently exceeding 150 minutes of at least moderate intensity exercise per week
* Report of chest pain, shortness of breath, fainting, or angina pectoris
* Self-reported history of falling, fall risk
* Have physical disability that would limit range of motion through exercises such as sitting, standing and inability to walk one block
* Plans to move from the area
* Enrolled in another clinical trial or has used of any investigational drugs, biologics, or devices within 30 days prior to study enrollment
* Self-reported tobacco use in last 7 days, current smoking, current tobacco use including e-cigarettes and vaping devices
* Not suitable for study participation due to other reasons at the discretion of the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Changes in Vascular Stiffness Following Distance-Based Exercise Program | 14 weeks
  Within participant change from pre- to post-intervention as measured by carotid-femoral pulse wave velocity, which is a measure of speed that is directly related to the stiffness of the arteries/vessels of the body.

SECONDARY OUTCOMES:
Changes in Vascular Function Following Distance-Based Exercise Program | 14 weeks
  Within participant change from pre- to post-intervention as measured by brachial artery time to flow mediated dilation, which is a measure of endothelial cell function responding to constriction and dilation of the arteries/vessels of the body. A faster FMD measure indicates better endothelial cell function, which indicates better vascular function.
Changes in Atherosclerotic Cardiovascular Disease (ASCVD) Risk Profiles Following a Distance-Based Exercise Program | 14 weeks
  Within participant change from pre- to post-intervention as measured by composite score expressed as a percentage from Atherosclerotic Cardiovascular Disease (ASCVD) Risk profile. ASCVD Risk score estimates the likelihood a person will develop atherosclerotic cardiovascular disease in the next 10 years. The higher the score, the more likely the person will have negative cardiovascular health outcomes. Less than 5% is considered a low score, and greater than 20% is considered a high score.

OTHER OUTCOMES:
Changes in Functional Fitness | 14 weeks
  Within participant change of functional fitness from pre- to post-intervention as measured by the Functional Fitness Test.
Estimation of Muscle Strengthening Exercise Session Adherence | 14 weeks
  Proportion of planned exercise sessions in which a participant completes at least 50% of prescribed exercises.
Estimation of Adherence to Aerobic Physical Activity Guidelines (150 minutes/week) | 14 weeks
  Proportion of planned weeks a participant accumulates 150 minutes of moderate intensity activity per week.
Estimation of Tele-Coaching Adherence | 14 weeks
  Proportion of planned coaching sessions in which a participant completes.
Estimation of Intervention Acceptability | 14 weeks
  Within participant change of questionnaire scores from pre- to post-intervention. Likert scale ratings of quality of exercise equipment, educational materials, health coaching, study feedback and distance delivery format. Five point Likert scale ranging from extremely dissatisfied/ important to extremely satisfied/important. I higher score shows more satisfaction or feeling of importance with study measures.
Change in Waist to Hip ratio (WHR) | 14 weeks
  Within participant changes of waist and hip circumference, expressed as the ratio of waist circumference relative to hip circumference from pre- to post-intervention. A waist to hip ratio of over 0.85 in women is higher risk for negative health outcomes.
Changes in body weight | 14 weeks
  Within participant changes of body weight from pre- to post-intervention.
Changes in Ambulatory Activity Levels | 2 weeks
  Within participant change in average daily steps taken within a week from pre- to post-intervention as measured via ActiGraph accelerometer.
Changes in self-efficacy relating to aerobic exercise | 14 weeks
  Within participant change of questionnaire scores from pre- to post-intervention. This questionnaire includes ten questions each with a score from 0-9, the questionnaire is scored by multiplying each question response by ten and then summing those values for a total score. Questionnaire ranges from 0-90 with a higher score indicating higher confidence (higher self efficacy) in the participant's ability to complete aerobic exercise.
Changes in self-efficacy relating to strength exercises | 14 weeks
  Within participant change of questionnaire scores from pre- to post-intervention. This questionnaire includes ten questions each with a score from 0-9, the questionnaire is scored by multiplying each question response by ten and then summing those values for a total score. Questionnaire ranges from 0-90 with a higher score indicating higher confidence (higher self efficacy) in the participant's ability to complete strength exercises.
Changes in the Basic Psychological Needs in Exercise Scale | 14 weeks
  Within participant change of questionnaire score from pre- to post-intervention. Eleven questions on a five-point Likert score from "I don't agree at all" to "I completely agree." This questionnaire is scored from 11 to 55 with 55 showing the most satisfaction with exercise. There are three subscales which include: autonomy, competence, and relatedness.
Changes in the Exercise Regulations Questionnaire | 14 weeks
  Within participant change of questionnaire score from pre- to post-intervention. This questionnaire includes 24 questions scored on a five-point Likert scale from "Not true for me" to "Very true for me" that is scored according to standard protocols taking composite measures of higher Likert ratings. Questionnaire scores range from 0-124 with a higher number indicating a higher engagement and regulations towards exercise.
Changes in the Multidimensional Scale of Perceived Social Support | 14 weeks
  Within participant change of questionnaire score from pre- to post-intervention. This questionnaire includes 12questions on a seven-point Likert scale with the lowest being "Very strongly disagree" to Very strongly agree" that is scored according to standard protocols taking composite measures of higher Likert rating. Questionnaire scores range from 12-84 with the higher number indicating more social support.
Changes in the Food Frequency Questionnaire | 14 weeks
  Within participant change of questionnaire score from pre- to post-intervention. This questionnaire includes 16 questions on a nine-point Likert scale from "Never" to "4 or more times per day." This questionnaire relates to the amount of food consumed, and that results are scored via categories of fat, protein, and fruits and vegetables. Questionnaire scores range from 0 to 128, with a higher number indicating higher consumption of dietary components.

CONTACTS AND LOCATIONS:
Overall Officials: Jess Gorzelitz, PHD, MS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT06534008/Prot_007.pdf
  • Informed Consent Form (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT06534008/ICF_008.pdf